CLINICAL TRIAL: NCT04125394
Title: Unicentric Clinical Trial on the Clinical Efficacy and Tolerance of the Treatment With an Ophthalmic Solution of Hypertonic Sodium Chloride (NaCl 5%) Without Preservatives in Patients Suffering From Symptomatic Corneal Edema
Brief Title: Efficacy and Tolerance of Hypertonic Sodium Chloride (NaCl 5%) Eye Drops Without Preservatives in Corneal Edema
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tiedra Farmacéutica SL (Industry)
Collaborators: Hospital Universitario Principe de Asturias (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCL/CSH/022019
Record Dates: First submitted 2019-10-11; First posted 2019-10-14 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Corneal Edema
Keywords: corneal edema; sodium chloride; single-dose
MeSH Terms: conditions — Corneal Edema

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NaCl 5% (Experimental): Hypertonic sodium chloride (NaCl 5%) eye drops solution in single-dose, without preservatives, administered every 8 hours for 28 days.
  Interventions: Device: hypertonic Sodium chloride (NaCl 5%) eye drops solution in single-dose

INTERVENTIONS:
Device: hypertonic Sodium chloride (NaCl 5%) eye drops solution in single-dose — Ophthalmic solution of hypertonic sodium chloride (NaCl 5%) without preservatives in single-dose container
  Other Names: Ocumax 5 eye drops solution in single-dose

SUMMARY:
Corneal edema is frequently found in clinical practice as a common sign of acute corneal disease due to different etiologies that cause an accumulation of extracellular fluid in the cornea. The present unicentric clinical trial aims to evaluate the efficacy and tolerance of an ophthalmic solution of hypertonic sodium chloride (NaCl 5%) without preservatives in participants suffering from symptomatic corneal edema.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Clinical diagnosis of symptomatic corneal edema related to chronic epithelial, secondary to corneal dystrophies, controlled infectious and inflammatory pathologies and surgical trauma already resolved.
* No need for keratoplasty in the 6 months following the start of the study

Exclusion Criteria:.

* Visual acuity less than 1/20 in both eyes
* Corneal edema caused by the following acute etiologies: trauma, infection, inflammation or Stevens-Johnson syndrome.
* Glaucoma or uncontrolled hypertension.
* Known allergy to any of the ingredients of the product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-02-03 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Mean Change from Baseline in Visual acuity | Baseline, Day 7 and Day 28

SECONDARY OUTCOMES:
Mean Change from Baseline in Corneal Thickness | Baseline, Day 7 and Day 28
  Micrometers

OTHER OUTCOMES:
Number of Participants with Treatment-Related Adverse Events (Objective Tolerance) | Baseline, Day 7 and Day 28
  Slit Lamp Examination
Score in Subjective Tolerance Test | Day 7 and Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Príncipe de Asturias, Alcalá de Henares, Spain

IPD SHARING:
Plan to Share IPD: Undecided